CLINICAL TRIAL: NCT05869799
Title: Effect of Vigiis 101 Lactic Acid Bacteria Powder on Body Weight and Body Fat in Overweight Participants: a Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Effect of Vigiis 101 Lactic Acid Bacteria Powder on Body Weight and Body Fat in Overweight Participants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SunWay Biotech Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24 Vigiis 101
Record Dates: First submitted 2023-03-15; First posted 2023-05-22 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Body Weight; Body Fat; Overweight
MeSH Terms: conditions — Body Weight; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This experiment adopts a block random assignment design, and the system assignment table (Block randomization, block size = 6) randomly generated by the program is given serial numbers and assigned to groups. The probability of assignment to each group is 1/2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vigiis 101 Lactobacillus Capsules (Experimental): Vigiis 101 Lactic Acid Bacteria Capsules is a commercially available product for Lactobacillus paracasei subspecies paracasei NTU 101 (NTU 101) is a strain of Lactobacillus isolated from the intestinal tract of newborns in Taiwan. 10 billion CFU/cap of NTU 101 freeze-dried powder (production research and development: Chenhui Biotechnology Co., Ltd. Biotechnology Co., Ltd., Taipei, Taiwan), corn starch, crystalline cellulose and excipients in vegetable capsules were prepared.
  Interventions: Dietary Supplement: Vigiis 101 Lactobacillus Capsules
- Placebo Capsules (Placebo Comparator): Maltodextrin was used as a placebo.
  Interventions: Dietary Supplement: Placebo Capsules

INTERVENTIONS:
Dietary Supplement: Vigiis 101 Lactobacillus Capsules — Product ingredients: microcrystalline cellulose, corn starch, NTU 101 lactic acid bacteria powder (1.0 x 10^10 CFU); capsule shell composition: HPMC (hydroxypropyl methylcellulose), purified water, titanium dioxide, gellan gum.
  Arms: Vigiis 101 Lactobacillus Capsules
Dietary Supplement: Placebo Capsules — Maltodextrin was used as a placebo
  Arms: Placebo Capsules

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, parallel-controlled trial (14 weeks in total), divided into three periods (screening, treatment, and discontinuation follow-up)

DETAILED DESCRIPTION:
Subjects meeting the inclusion criteria were randomly assigned to 2 groups (Vigiis 101 lactic acid bacteria: n = 50, placebo: n = 50) in a 1:1 ratio, Block : 4 randomization. Randomization was performed by a research statistician not directly involved in the trial. Researchers and subjects were unaware of treatment groups until data analysis was complete.

During the 12-week use trial, subjects were asked to take Vigiis 101 Lactobacillus capsules or a placebo once a day before breakfast. The subjects were required to maintain a regular lifestyle and recorded daily Vigiis 101 Lactobacillus or placebo consumption, diet and the number of steps walked as a measure of physical activity. Body composition, anthropometric and biochemical measurements were measured at weeks 0, 4, 8, and 12 after consumption initiation. Clinical exams are done every 4 weeks in the hospital. Subjects filled out daily diaries that included questions about study product intake, other food intake, number of bowel movements, stool quality (consistency and color), any medications received, and any uncomfortable symptoms such as diarrhea, constipation, Vomiting, flatulence, discomfort, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are 20-65-year-old men or non-pregnant women (women of childbearing age are not allowed to become pregnant or breastfeed during the study) and adult volunteers who are conscious and able to communicate.
2. Subjects with a body mass index (BMI) between 23 and 29.9 (kg/m2 ) and classified as overweight according to the World Health Organization Asia-Pacific criteria.
3. Subjects who agree to participate in this trial and voluntarily agree to the test consent in writing.

Exclusion Criteria:

1. Subjects who are pregnant or lactating or expecting pregnancy.
2. Those with gallbladder disease, gastrointestinal disease, gout, porphyria (Porphyria) or a history of stomach weight control surgery.
3. Subjects suffering from high blood pressure (≥160/100 mmHg, after resting for 10 minutes) or taking diuretics.
4. Subjects with diabetes (fasting blood glucose (≥125 mg/dL).
5. Suffering from heart disease, liver and kidney insufficiency, hyperthyroidism or hypothyroidism, Cushing's syndrome, malignant tumor or any other diseases that affect the research results.
6. Suffering from depression, schizophrenia, alcoholism, drug addiction and other mental disorders or taking drugs (such as psychotropic drugs, β receptor blockers).
7. Subjects have taken drugs that may affect body weight or body fat (such as contraceptives, steroids, female hormones) or functional foods within 2 weeks before the screening visit.
8. Subjects judged to be unable to exercise due to severe musculoskeletal diseases.
9. Subjects who consumed probiotics or expected to consume probiotics within 2 weeks before the screening visit.
10. Subjects who have participated in or are expected to participate in clinical trials within 4 weeks before the screening visit.

The withdrawal criteria are as follows:

(1) Unable to take the test sample on time (i.e. more than 7 days out of every 4 weeks without taking the sample) (2) Unable to cooperate with the return visit on time (after being contacted or lost contact, 7 days beyond the expected return visit time) (2) If the subject chooses to voluntarily stop participating due to personal reasons.

(3) Serious violations of the research protocol. (4) Taking drugs that may affect body weight or body fat (such as contraceptives, steroids, female hormones) or functional health food with probiotics in the experiment.

(5) When severe adverse reactions occur clinically. (6) The aforementioned "subject exclusion conditions" did not occur during the screening period, and must be withdrawn if they occur during the trial.

(7) Other situations where continuing to participate in the research will endanger the health of the subject. When there is important new information during the execution of the trial (referring to your rights or affecting your willingness to continue participating), you will be notified and further explained. Please reconsider whether to continue participating. You can decide freely and will not cause any discomfort. Or affect their future physicians to your medical care.

(8) The project host or the sponsor may also suspend the entire experiment if necessary.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
BMI improvement | 12 weeks
  Improvement in BMI from baseline was used as the primary outcome.

SECONDARY OUTCOMES:
Other body index improvements | 12 weeks
  The secondary outcome was the improvement in body fat percentage (measured in %).

CONTACTS AND LOCATIONS:
Overall Officials: WEN-HUI FANG, Ph. D., Principal Investigator — Chief of Family medicine department
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Breton J, Galmiche M, Dechelotte P. Dysbiotic Gut Bacteria in Obesity: An Overview of the Metabolic Mechanisms and Therapeutic Perspectives of Next-Generation Probiotics. Microorganisms. 2022 Feb 16;10(2):452. doi: 10.3390/microorganisms10020452. PMID 35208906
- [Result] Chiang SS, Pan TM. Antiosteoporotic effects of Lactobacillus -fermented soy skim milk on bone mineral density and the microstructure of femoral bone in ovariectomized mice. J Agric Food Chem. 2011 Jul 27;59(14):7734-42. doi: 10.1021/jf2013716. Epub 2011 Jun 21. PMID 21668014
- [Result] Chiu CH, Lu TY, Tseng YY, Pan TM. The effects of Lactobacillus-fermented milk on lipid metabolism in hamsters fed on high-cholesterol diet. Appl Microbiol Biotechnol. 2006 Jun;71(2):238-45. doi: 10.1007/s00253-005-0145-0. Epub 2005 Sep 20. PMID 16172889
- [Result] Cheng MC, Tsai TY, Pan TM. Anti-obesity activity of the water extract of Lactobacillus paracasei subsp. paracasei NTU 101 fermented soy milk products. Food Funct. 2015 Nov;6(11):3522-30. doi: 10.1039/c5fo00531k. Epub 2015 Aug 24. PMID 26299532
- [Result] Leon Aguilera XE, Manzano A, Pirela D, Bermudez V. Probiotics and Gut Microbiota in Obesity: Myths and Realities of a New Health Revolution. J Pers Med. 2022 Aug 4;12(8):1282. doi: 10.3390/jpm12081282. PMID 36013231
- [Result] Liu CF, Tung YT, Wu CL, Lee BH, Hsu WH, Pan TM. Antihypertensive effects of Lactobacillus-fermented milk orally administered to spontaneously hypertensive rats. J Agric Food Chem. 2011 May 11;59(9):4537-43. doi: 10.1021/jf104985v. Epub 2011 Apr 4. PMID 21446645
- [Result] Liu TH, Tsai TY, Pan TM. The Anti-Periodontitis Effects of Ethanol Extract Prepared Using Lactobacillus paracasei subsp. paracasei NTU 101. Nutrients. 2018 Apr 12;10(4):472. doi: 10.3390/nu10040472. PMID 29649103
- [Result] Musazadeh V, Zarezadeh M, Ghalichi F, Ahrabi SS, Jamilian P, Jamilian P, Ghoreishi Z. Anti-obesity properties of probiotics; a considerable medical nutrition intervention: Findings from an umbrella meta-analysis. Eur J Pharmacol. 2022 Aug 5;928:175069. doi: 10.1016/j.ejphar.2022.175069. Epub 2022 Jun 1. PMID 35659967
- [Result] Nam GE, Kim YH, Han K, Jung JH, Rhee EJ, Lee WY; Obesity Fact Sheet of the Korean Society for the Study of Obesity. Obesity Fact Sheet in Korea, 2020: Prevalence of Obesity by Obesity Class from 2009 to 2018. J Obes Metab Syndr. 2021 Jun 30;30(2):141-148. doi: 10.7570/jomes21056. PMID 34158420
- [Result] Ridaura VK, Faith JJ, Rey FE, Cheng J, Duncan AE, Kau AL, Griffin NW, Lombard V, Henrissat B, Bain JR, Muehlbauer MJ, Ilkayeva O, Semenkovich CF, Funai K, Hayashi DK, Lyle BJ, Martini MC, Ursell LK, Clemente JC, Van Treuren W, Walters WA, Knight R, Newgard CB, Heath AC, Gordon JI. Gut microbiota from twins discordant for obesity modulate metabolism in mice. Science. 2013 Sep 6;341(6150):1241214. doi: 10.1126/science.1241214. PMID 24009397
- [Result] Tsai TY, Chu LH, Lee CL, Pan TM. Atherosclerosis-preventing activity of lactic acid bacteria-fermented milk-soymilk supplemented with Momordica charantia. J Agric Food Chem. 2009 Mar 11;57(5):2065-71. doi: 10.1021/jf802936c. PMID 19216552
- [Result] Tsai YT, Cheng PC, Pan TM. Immunomodulating activity of Lactobacillus paracasei subsp. paracasei NTU 101 in enterohemorrhagic Escherichia coli O157H7-infected mice. J Agric Food Chem. 2010 Nov 10;58(21):11265-72. doi: 10.1021/jf103011z. Epub 2010 Oct 13. PMID 20942489
- [Result] Tsai YT, Cheng PC, Fan CK, Pan TM. Time-dependent persistence of enhanced immune response by a potential probiotic strain Lactobacillus paracasei subsp. paracasei NTU 101. Int J Food Microbiol. 2008 Dec 10;128(2):219-25. doi: 10.1016/j.ijfoodmicro.2008.08.009. Epub 2008 Aug 26. PMID 18809220
- [Result] Vallianou N, Dalamaga M, Stratigou T, Karampela I, Tsigalou C. Do Antibiotics Cause Obesity Through Long-term Alterations in the Gut Microbiome? A Review of Current Evidence. Curr Obes Rep. 2021 Sep;10(3):244-262. doi: 10.1007/s13679-021-00438-w. Epub 2021 May 4. PMID 33945146